CLINICAL TRIAL: NCT04107493
Title: Evaluation of a Portable Oxygen Concentrator During Ambulation for Patients Who Require Supplemental Oxygen (POC-LEAN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MA-19-03-02
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, cross-over study design with participants serving as their own controls. A within- participants, repeated-measures design is used during 6MWT. Eligible participants will complete two 6MWTs: one with their usual portable oxygen cylinder, and one with Mobi™. All participants entered into the study will be randomized in a 1:1 ratio to the following order of device use:
  * Control device (portable oxygen cylinder) first; or
  * Study device (Mobi™, POC) first.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Portable oxygen cylinder (Active Comparator): Continuous flow oxygen cylinders will be used as a comparison.
  Interventions: Device: Portable Oxygen Cylinder
- Mobi™ Portable Oxygen Concentrator (Experimental): Mobi™ is indicated for patients who require supplemental oxygen, including COPD patients. It provides supplemental, high oxygen concentration to these patients. It is available via prescription only and may be used in the home, institution, and hospital settings, as well as travel environments
  Interventions: Device: Mobi

INTERVENTIONS:
Device: Portable Oxygen Cylinder — A POC is a medical device that is indicated for patients who require supplemental oxygen, including COPD patients
  Other Names: POC
  Arms: Portable oxygen cylinder
Device: Mobi — ResMed's variant of POC
  Other Names: Mobi POC
  Arms: Mobi™ Portable Oxygen Concentrator

SUMMARY:
Prospective randomized study with a cross-over design. Mobi™ is a relatively new POC in the market and thus it is valuable to collect data from COPD patients using supplemental oxygen, and their use on Mobi™. The purpose of the present study is to compare Mobi™ with a continuous flow oxygen cylinder, with SpO2 as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. Male or female, age ≥ 18 years at the time of signing informed consent.
3. Diagnosed with COPD and currently in a stable state (at least 4 weeks since last exacerbation episode22).
4. Current prescription for long-term oxygen therapy.
5. Participants meet the criteria for pulse-dose portable oxygen delivery, defined as being mobile within the home and the qualifying blood gas study was performed at rest/ awake or during exercise.
6. Participants who can read and comprehend English.

Exclusion Criteria:

1. Clinically unstable, in the investigator's opinion, which might jeopardize the participant's safety or compliance with the protocol.
2. Current oxygen therapy prescription for >5 L/min continuous flow.
3. Known or suspected contraindication for pulse-dose oxygen.
4. Unable to complete 6MWTs, e.g., unstable angina and myocardial infarction during the previous month
5. Female who is pregnant, breast-feeding, or intends to become pregnant, or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Clark, M.D, Principal Investigator — SleepData
Locations (1):
- SleepData, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gloeckl R, Jarosch I, Schneeberger T, Fiedler C, Lausen M, Weingaertner J, Hitzl W, Kenn K, Koczulla AR. Comparison of supplemental oxygen delivery by continuous versus demand based flow systems in hypoxemic COPD patients - A randomized, single-blinded cross-over study. Respir Med. 2019 Sep;156:26-32. doi: 10.1016/j.rmed.2019.08.001. Epub 2019 Aug 5. PMID 31404750
- [Background] Guell Rous R. Long-term oxygen therapy: are we prescribing appropriately? Int J Chron Obstruct Pulmon Dis. 2008;3(2):231-7. doi: 10.2147/copd.s1230. PMID 18686732

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants acted as their own controls. Participants were randomised as to the order they used the devices during the 6-minute walking test. There was a one hour wash out period between tests
Groups:
- Portable Oxygen Cylinder, Then Mobi; Mobi, Then Portable Oxygen Cylinder: Participants acted as their own control in this study.
  Participants used two portable oxygen cylinders during a 6 minute walk test. One was a standard POC, and one was the trial device, the Mobi POC
  Portable Oxygen Cylinder: A POC is a medical device that is indicated for patients who require supplemental oxygen, including COPD patients
Period: First Intervention (1 Hour)
Arm/Group | Portable Oxygen Cylinder, Then Mobi | Mobi, Then Portable Oxygen Cylinder
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: Washout (One Hour)
Arm/Group | Portable Oxygen Cylinder, Then Mobi | Mobi, Then Portable Oxygen Cylinder
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Portable Oxygen Cylinder, Then Mobi | Mobi, Then Portable Oxygen Cylinder
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: COPD adult patients with long term oxygen therapy history were included. They were all stable (at least 4 weeks since last exacerbation episode).
Groups:
- All Study Participants: Participants acted as their own control during this study. Participants used a portable oxygen cylinder whilst doing a 6 minute walking test. After a wash out period the participants completed the 6 minute walking test with the second portable oxygen cylinder. The order of the oxygen cylinders (mobi or standard) was randomised
Arm/Group | All Study Participants
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.86 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean SpO2 (Oxygen Saturation) During Six Minute Walk Tests (6MWTs)
Description: Each subject's SpO2 will be measured when each subject takes six minutes walk test
Time Frame: Mean Sp02, measured during 6 minute walk test
Measure: Mean (Standard Error); unit: percentage of oxygen saturation
Arm/Group | Portable Oxygen Cylinder | Mobi™ Portable Oxygen Concentrator
Number analyzed (Participants) | 33 | 33
percentage of oxygen saturation | 91.2 (0.7) | 90.0 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the one study visit. After completion of this visit, the participants involvement in the study was completed
Groups:
- Standard Oxygen Cylinder; Mobi: Participants acted as their own control in this study.
  Participants used two portable oxygen cylinders during a 6 minute walk test. One was a standard POC, and one was the trial device, the Mobi POC
  Portable Oxygen Cylinder: A POC is a medical device that is indicated for patients who require supplemental oxygen, including COPD patients
Arm/Group | Standard Oxygen Cylinder | Mobi
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT04107493/Prot_SAP_000.pdf